CLINICAL TRIAL: NCT03536455
Title: Effect of Acetazolamide on Maximal Exercise Performance in Lowlanders Older Than 40 Years at Altitude: A Randomized, Placebo-controlled, Double-blind Parallel Trial
Brief Title: Effect of Acetazolamide on Maximal Exercise Performance in Lowlanders Older Than 40 Years at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-01-8/305B
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Altitude Hypoxia
Keywords: healthy participants older than 40 years; exercise performance; prevention; acetazolamide
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 1x125mg acetazolamide in the morning, 2x125mg in the evening, starting 24 hours before departure to 3'100m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3'100m
  Arms: PLACEBO oral capsule

SUMMARY:
Randomized, placebo controlled trial evaluating the effect of acetazolamide on maximal exercise performance in lowlanders older than 40 years travelling from 760 m to 3'100 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the effect of acetazolamide intake on the maximal exercise performance in lowlanders older than 40 years travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3'100 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo), will be administered before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3'100 m.

An interim analysis will be carried out when 80 participants will have completed the study or after the first year. The Peto's method will be used and the trial will be stopped when pre-specified futility boundaries were crossed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, age 40-75 yrs, without any disease and need of medication.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.
* Kyrgyz ethnicity

Exclusion Criteria:

* Any active respiratory, cardiovascular or other disease requiring regular treatment or being otherwise relevant for tolerance of hypoxia or altitude exposure.
* Any condition that may interfere with protocol compliance including current heavy smoking (>20 cigarettes per day or >20 pack-years with active smoking during the last 10 years), regular use of alcohol.
* Allergy to acetazolamide and other sulfonamides.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Change in maximal power output during exercise | Day 1 at 760m and day 1 at 3'100m
  Difference in altitude-induced change in maximal power output between acetazolamide and placebo group.

SECONDARY OUTCOMES:
Change in peak oxygen uptake during exercise | Day 1 at 760m and day 1 at 3'100m
  Difference in altitude-induced change in peak oxygen uptake between acetazolamide and placebo group.
Change in cerebral tissue oxygenation during exercise | Day 1 at 760m and day 1 at 3'100m
  Difference in altitude-induced change in cerebral tissue oxygenation between acetazolamide and placebo, measured by near-infrared spectroscopy during cycle spiroergometry
Change in muscle tissue oxygenation during exercise | Day 1 at 760m and day 1 at 3'100m
  Difference in altitude-induced change in muscular tissue oxygenation between acetazolamide and placebo, measured by near-infrared spectroscopy during cycle spiroergometry
Change in arterial blood gasses at rest and peak exercise | Day 1 at 760m and day 1 at 3'100m
  Difference in altitude-induced change in arterial blood gases between acetazolamide and placebo measured before and at peak exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan; Michael Furian, MSc, Principal Investigator — University Hospital, Zürich
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan